CLINICAL TRIAL: NCT01903564
Title: Fetal and Neonatal Magnetophysiology
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Shared Medical Technology, Inc. (Industry); Medical College of Wisconsin (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2013-0362; R01HL063174 (NIH)
Record Dates: First submitted 2013-07-11; First posted 2013-07-19 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Fetal Arrhythmia; Abnormality in Fetal Heart Rate or Rhythm; Long QT Syndrome
Keywords: fetus; fetal arrhythmia; fetal heart rate; long QT syndrome
MeSH Terms: conditions — Long QT Syndrome | interventions — Magnetocardiography; Electrocardiography; Ultrasonography, Doppler; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normal: pregnant women with uncomplicated pregnancies
  Interventions: Device: magnetocardiography; Device: fetal echocardiography
- high-risk: pregnant women with pregnancies complicated by fetal arrhythmia or the risk of fetal arrhythmia
  Interventions: Device: magnetocardiography; Device: postnatal ECG; Device: fetal echocardiography

INTERVENTIONS:
Device: magnetocardiography — recording of magnetic heart activity
  Other Names: MCG; fetal magnetocardiography
Device: postnatal ECG — postnatal ECG
  Other Names: electrocardiography
  Groups: high-risk
Device: fetal echocardiography — fetal echocardiography
  Other Names: Doppler ultrasound; M-mode ultrasound; 2d ultrasound

SUMMARY:
Fetal research and clinical practice has been hampered by a lack of suitable investigational techniques. Currently, ultrasound is the only widely used method of studying fetal anatomy and physiology, but it has significant limitations for assessment of cardiac rhythm. The proposed study will allow us to investigate fetal magnetocardiography (fMCG) as a new tool for the study of normal and abnormal fetal heart rate and rhythm, with a goal of demonstrating probable benefit from use of the device in patients with serious fetal arrhythmia. We propose a study that will last 1-2 years and will provide data to aid in assessing the safety and effectiveness of fMCG for diagnosis and management of patients with abnormal fetal heart rate and rhythm. We hope that the data from the study will support a Humanitarian Device Exemption (HDE) application for the subject device. The safety and efficacy study designs are described below. High-risk subjects will undergo echocardiography as part of their routine clinical management, and our results will be compared to the echocardiography results, as well as with postnatal ECG, when available. (Since many arrhythmias resolve prior to birth, either due to resolution of disease or due to treatment, only a limited number of diseases allow postnatal comparison). For rhythms that persist after birth, the diagnostic utility of fMCG and echocardiography will be assessed by computing the sensitivity (Sn) and specificity (Sp) relative to postnatal ECG for the following prenatal modalities: (i) the fMCG, (ii) the original (referral) echo, (iii) if available, the in-lab echocardiogram at the time of the fMCG study. Secondary endpoints will assess changes in diagnosis and in clinical management due to the additional information provided by fMCG, compared to the information provided by echocardiography alone.

ELIGIBILITY:
Inclusion Criteria:

Normal subjects: normal, healthy adult women with uncomplicated pregnancies

High-risk cohort: The primary inclusion criterion is diagnosis of serious fetal arrhythmia, which is defined as sustained low or high heart rate. Low heart rate, or bradycardia, and high heart rate, or tachycardia, are based on normative values for gestation (usually below 110 -120 beats/min, or above 160-180 beats/min). Intermittent bradycardia and tachycardia are also important to detect because these arrhythmias may become incessant over the course of pregnancy and have implications for patient management. Abnormal repolarization, such as long QT syndrome (LQTS), is another important class of arrhythmia. Fetuses with a family history of LQTS or a suspicious rhythm (low heart rate, intermittent AV block, or ventricular tachycardia) will also be studied.

Exclusion Criteria:

The pregnant women subjects must by aged 18 or older. High-risk subjects cannot participate if their physician in consultation with the lead physician of the study does not grant permission for them to participate in the study due to risk of travel or other reason.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We plan to study a total of 180 subjects. Sixty will be pregnant women with uncomplicated pregnancies; 120 will be pregnant women with pregnancies complicated by fetal arrhythmia or a condition that puts the fetus at risk of fetal arrhythmia. We refer to these cases as "high-risk" due to the presence of or risk of arrhythmia to the fetus. The pregnant mothers will be age 18 or older. They will be studied as early as 15 weeks' gestation and may be asked to return, if their physician determines that additional fMCG studies are necessary.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wakai, Ph.D., Principal Investigator — University of Wisconsin, Madison; Janette Strasburger, M.D., Study Director — Medical College of Wisconsin
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal | High-risk
Started | 10 | 29
Completed | 10 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal | High-risk | Total
Number analyzed (Participants) | 10 | 29 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 29 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 31.8 [28 to 35] | 32.0 [24 to 42] | 31.9 [24 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 29 | 39
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 29 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Experiencing Symptoms
Description: Percentage of subjects experiencing symptoms
Time Frame: 15-40 weeks' gestation
Population: Symptoms include premature labor, vaginal bleeding, uterine cramping, nausea/vomiting, dizziness, dsypnea, syncope, palpitations, or fatigue during the study session.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal | High-risk
Number analyzed (Participants) | 10 | 29
Participants | 0 | 0

2. Primary Outcome: Percentage of Subjects Experiencing Adverse Events Unrelated to Device
Description: Percentage of subjects experiencing adverse events unrelated to device
Time Frame: 15 weeks' gestation till up to 1 month after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Normal | High-risk
Number analyzed (Participants) | 10 | 29
Participants | 0 | 10

3. Primary Outcome: Number of Participants With Concordance of fMCG and Postnatal ECG for Diagnosis of Long QT Syndrome
Description: Number of Participants with Concordance of fMCG and Postnatal ECG for Diagnosis of Long QT Syndrome based on measurement of rate-corrected QT interval (QTc)
Time Frame: Birth to age 1 week
Population: Fetuses with a family history of long QT syndrome
Measure: Count of Participants; unit: Participants
Arm/Group | Normal | High-risk
Number analyzed (Participants) | 0 | 6
Participants | 0 | 6

4. Primary Outcome: Percentage of Subjects Experiencing Adverse Events Related to Device
Description: Percentage of Subjects Experiencing Adverse Events Related to Device
Time Frame: 15 weeks' gestation till up to 1 month after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Normal | High-risk
Number analyzed (Participants) | 10 | 29
Participants | 0 | 0

5. Secondary Outcome: Percentage of Fetuses With a Family History of Long QT Syndrome Who a Change in Diagnosis Due to fMCG
Description: Percentage of fetuses with a family history of long QT syndrome who a change in diagnosis due to fMCG
Time Frame: 15 weeks' gestation to birth
Population: Fetuses with family history of LQTS
Measure: Count of Participants; unit: Participants
Arm/Group | Normal | High-risk
Number analyzed (Participants) | 0 | 6
Participants | 0 | 3

6. Secondary Outcome: Percentage of Fetuses With a Family History of Long QT Syndrome Who Had a Change in Management Due to fMCG
Description: Percentage of fetuses with a family history of long QT syndrome who had a change in management due to fMCG
Time Frame: 15 weeks' gestation to birth
Population: Fetuses with a family history of fetal long QT syndrome
Measure: Count of Participants; unit: Participants
Arm/Group | Normal | High-risk
Number analyzed (Participants) | 0 | 6
Participants | 0 | 2

ADVERSE EVENTS:
Arm/Group | Normal | High-risk
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/29
Other Adverse Events (participants affected / at risk) | 0/10 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal (N=10) | High-risk (N=29)
fetal death (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — A fetus with a severe ion channelopathy died 10 days following participation in the study. The death is believed to be unrelated to the use of the device.
Motor vehicle accident (General disorders) | 0 (0) | 1 (1) — Subject was driving and was rear ended at high speed by another car. OB chose to admit her over night for observation for possibility of uterine contractions. No problem in-house, sent home <24 hours later.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No